CLINICAL TRIAL: NCT03826134
Title: Interventional, Phase I, Open-label, First in Human, Single-center Positron Emission Tomography (PET) Study Investigating Test-retest Properties of [11C]-PXT012253 as a Radiotracer in Healthy Subjects
Brief Title: A Positron Emission Tomography (PET) Study to Examine the Brain Binding Properties of a Novel Radioactive Compound [11C]-PXT012253 in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18039A
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [11C]-PXT012253 (Experimental)
  Interventions: Drug: [11C]PXT012253

INTERVENTIONS:
Drug: [11C]PXT012253 — Single intravenous bolus injection. The injected amount will be less than 5 μg. The radioactive dose is approximately 400 MBq per 70 kg body weight.

SUMMARY:
This study evaluates the usefulness of a PET radioligand to estimate the binding on the mGlu4 receptor in the brain. mGlu4 has been proposed as a therapeutic target in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects age 20-50 inclusive
* Body mass index (BMI) between 19 and 30 kg/m2
* Normal sMRI scan, performed within 3 months, as judged by the investigator
* The subject is, in the opinion of the investigator, generally healthy based on assessment of medical history, physical examination, vital signs, ECG, and the results of the hematology, clinical chemistry, urinalysis, serology, and other laboratory tests
* Women of childbearing potential and men whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial and for 3 months thereafter
* A propensity to tolerate confined spaces for prolonged periods
* Suitability for radial and/or brachial artery blood sampling and cannulation

Exclusion Criteria:

* History of clinically significant cardio-or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder or any other major disorder that may interfere with the objectives of the study, as judged by the investigator
* The subject has 1 or more clinical laboratory test values outside the reference range, which in the opinion of the investigator are clinically significant
* Screening supine blood pressure >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility
* The subject has a resting pulse <=50 or >=100 bpm at the Screening Visit
* The subject has a QTc interval >430 ms (Bazett's or Fridericia's correction) at the Screening Visit or at he Baseline Visit, as calculated by the ECG equipment and evaluated by the investigator. The ECG may be repeated if any of the values are out-of-range or abnormal
* The subject is pregnant or breastfeeding
* Habitual use of nicotine products and addictive substances
* Any finding of significance on MRI scans as judged by the investigator.
* Any previous PET measurements for scientific purposes
* Use of CNS active drugs and/or NSAIDs 1 month prior to the first PET examination
* The subject is exposed to significant level of ionizing radiation at work
* The subject has undergone any clinical procedures involving significant exposure to radiation (excluding dental X-ray and common X-rays of the chest or extremities)
* The subject has received radio labeled material less than 12

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Total distribution volumes (VT) for each region of interest (ROI) | Up to 3 days
Binding potential (BPND) in the ROI's | Up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Karolinska Institute, Dept. of Clinical Neuroscience, Stockholm, Sweden